CLINICAL TRIAL: NCT04902222
Title: Incidence of Orthostatic Intolerance and Orthostatic Hypotension After Administration of Intravenous Morphine in Patients Prior to Hip or Knee Arthroplasty
Brief Title: Orthostatic Intolerance and Hypotension After Administration of Morphine in Patients Prior to Hip or Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Kehlet, Henrik, M.D., Ph.D. (Individual)
Responsible Party: Principal Investigator, Bodil Uldall-Hansen, Research assistant, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-20071567
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Orthostatic Hypotension; Orthostatic Intolerance
Keywords: Orthostatic Hypotension; Orthostatic Intolerance; Morphine; Autonomic Dysfunction
MeSH Terms: conditions — Hypotension, Orthostatic; Orthostatic Intolerance; Primary Dysautonomias | interventions — Morphine; Analgesics, Opioid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing primary hip or knee arthroplasty: Patients undergoing primary hip or knee arthroplasty
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Administration of 0.1 mg/kg (IBW) intravenous morphine
  Other Names: opioid

SUMMARY:
Incidence of orthostatic intolerance and orthostatic hypotension after intravenous administration of morphine in patients prior to hip or knee arthroplasty.

DETAILED DESCRIPTION:
Early postoperative mobilization is crucial for recovery of patients undergoing surgery in the multimodal fast-track approach to perioperative care, since physical immobilization is highly associated with increased risk of postoperative complications and prolonged hospital length of stay. Postoperative mobilization is often delayed due to patients experiencing orthostatic hypotension (OH), defined as a drop in systolic blood pressure > 20 mmHg or diastolic blood pressure > 10 mmHg, or orthostatic intolerance (OI), characterized by dizziness, blurred vision, nausea, vomiting, sensation of heat or syncope.

Previous studies have found a high incidence of postoperative OI (> 40 %) among patients undergoing total hip arthroplasty.

A possible causative factor to the high occurrence of OH and OI after surgery could be postoperative pain management by administration of morphine. Morphine is known to have many side-effects including nausea, vomiting, dizziness and orthostatic hypotension.

The object of this study is to isolate and estimate the effect of intravenous morphine on the incidence of OH and OI.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary unilateral total hip arthroplasty (THA), total knee arthroplasty (TKA) or unicompartmental knee arthroplasty (UKA)
* Patients > 18
* Patients that understand and speak Danish
* Patients that have provided written informed consent

Exclusion Criteria:

* Alcohol or substance abuse
* Habitual use of opioids
* Habitual use of anxiolytic, antidepressant and/or antipsychotic drugs
* History of previous orthostatic intolerance or hypotension
* Cognitive dysfunction
* Glomerular filtration rate (GFR) < 30 ml/min
* Cardiac arrhythmia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary unilateral total hip arthroplasty, total knee arthroplasty or unicompartmental knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of orthostatic hypotension | 30 minutes after morphine administration
  Orthostatic hypotension is defined as a fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg during mobilization

SECONDARY OUTCOMES:
Changes in systolic arterial pressure (SAP) during mobilization | Before and 30 minutes after morphine administration
  Measured in mmHg by non-invasive Lithium Dilution Cardiac Output (LiDCO) measurement
Changes in diastolic arterial pressure (DAP) during mobilization | Before and 30 minutes after morphine administration
  Measured in mmHg by non-invasive LiDCO
Changes in mean arterial pressure (MAP) during mobilization | Before and 30 minutes after morphine administration
  Measured in mmHg by non-invasive LiDCO
Changes in heart rate (HR) during mobilization | Before and 30 minutes after morphine administration
  Measured in beats min-1 by non-invasive LiDCO
Changes in stroke volume (SV) during mobilization | Before and 30 minutes after morphine administration
  Measured in mL by non-invasive LiDCO
Changes in cardiac output (CO) during mobilization | Before and 30 minutes after morphine administration
  Measured in L/min by non-invasive LiDCO
Changes in systemic vascular resistance (SVR) during mobilization | Before and 30 minutes after morphine administration
  Measured in dynes s cm-5 by non-invasive LiDCO
Changes in peripheral perfusion index (PPI) during mobilization | Before and 30 minutes after morphine administration
  Measured in % by Root Masimo
Changes in cerebral perfusion (ScO2) during mobilization | Before and 30 minutes after morphine administration
  Measured in % by Root Masimo
Changes in muscular perfusion (SmO2) during mobilization | Before and 30 minutes after morphine administration
  Measured in % by Root Masimo
Changes in baroreflex sensitivity - vagal (BRSv) during Valsalva manoeuvre | Before and 30 minutes after morphine administration
  Measured in ms
Changes in heart rate variability (HRV) during Valsalva manoeuvre | Before and 30 minutes after morphine administration
  Measured in ms

OTHER OUTCOMES:
Pain score during mobilisation | Before and 30 minutes after morphine administration
  Measured by verbal rating scale (VRS) from 0 to 10 (0 = no pain, 10 = worse pain imaginable)
Occurence of side-effects to morphine administration | 30 minutes after morphine administration
  Occurrence of following side-effects to morphine administration: nausea, vomiting, pruritus, headache or dizziness

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Bang Foss, Dr. Med., Study Director — Copenhagen University Hospital, Hvidovre
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No